CLINICAL TRIAL: NCT01278316
Title: Remote Administration Of Cognitive Training Tasks In Rural Veterans With PTSD And Comorbid Mild TBI: A Feasibility Study
Brief Title: Rural Veterans With Post-traumatic Stress Disorder (PTSD) And Comorbid Mild Traumatic Brain Injury (TBI): A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: South Central VA Mental Illness Research, Education & Clinical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mary Newsome, PI, Michael E. DeBakey VA Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-27735; 10K09.H (Other: MEDVAMC Research & Development Board)
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Post-Traumatic Stress Disorders; Traumatic Brain Injury
Keywords: PTSD; TBI; Cognition; Cognitive Training
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive training (Experimental): Cognitive Intervention Tasks Participants will be asked to perform the Brain Fitness (PositScience) cognitive training tasks an hour each day, five days per week for 8-10 weeks. Six tasks manipulating auditory and verbal information will be presented, and stimuli from all tasks are presented auditorily. All tasks are designed to begin with the lowest level of difficulty required to attain 85% accuracy, and as performance improves, difficulty increases to maintain 85% accuracy, with difficulty decreasing if accuracy decreases.
  Interventions: Behavioral: Cognitive Training
- Control (Active Comparator): The control group will perform computerized tasks that utilize cognitive performance, but were not systematically developed to improve cognitive performance.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Control — Participants will be asked to perform computerized tasks that involve auditory and verbal performance one hour each day, five days per week for 8-10 weeks. Six tasks requiring auditory and verbal information will be presented.
  Arms: Control
Behavioral: Cognitive Training — Participants will be asked to perform the Brain Fitness (PositScience) cognitive training tasks an hour each day, five days per week for 8-10 weeks. Six tasks manipulating auditory and verbal information will be presented, and stimuli from all tasks are presented auditorily. All tasks are designed to begin with the lowest level of difficulty required to attain 85% accuracy, and as performance improves, difficulty increases to maintain 85% accuracy, with difficulty decreasing if accuracy decreases.
  Arms: Cognitive training

SUMMARY:
This study is being conducted to understand whether training in tasks that require perceiving and thinking about things, or cognition, can improve memory in veterans who have been exposed to a blast explosion and have TBI and PTSD. A primary goal of the study is to determine whether it is feasible for veterans who don't live close to a VA to perform this cognitive training at home.

DETAILED DESCRIPTION:
Many military personnel have experienced traumatic brain injury (TBI) and posttraumatic stress disorder (PTSD) as a result of the current Afghanistan and Iraq wars. TBI occurs when a sudden force causes the brain to move, causing damage to brain cells. PTSD is an anxiety disorder associated with serious traumatic events. Blast explosions can lead to TBI. People who experience TBI as a result of a blast injury are more likely to experience PTSD than people who have TBI not due to blast. TBI and PTSD may be associated with memory problems in some patients. Because therapy for PTSD sometimes requires learning new ways to think about things and making new responses, being able to remember the new information being learned is important. It is possible that improving memory may also improve PTSD treatment.

This is a prospective study of Operation Enduring Freedom and Operation Iraqi Freedom (Afghanistan and Iraq wars; OEF/OIF) veterans who will undergo two neuropsychological and psychiatric assessments prior and subsequent to a cognitive training intervention. This is a feasibility study to ascertain whether OEF/OIF veterans diagnosed with mild TBI and comorbid PTSD and who live in rural locations will adhere to the schedule demands required of a computer-based cognitive training protocol.

ELIGIBILITY:
Inclusion Criteria:

* Rural residence
* Willingness to commit to the time requirements of the study
* Undergoing treatment for posttraumatic stress disorder (PTSD) as assessed by a clinician, diagnosed with mild traumatic brain injury (TBI)
* Native English speaker
* 20-40 years
* Normal or corrected to normal vision and hearing.

Exclusion Criteria:

* Substance dependence
* Major depression with suicidal ideation
* Psychotic disorder
* History of neurological disorder other than mild traumatic brain injury (TBI) due to blast from Operation Enduring Freedom (OEF) and Operation Iraqi Freedom (OIF) (i.e., Afghanistan and Iraq wars) deployment
* History of known or suspected learning disorder.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-01; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Compliance rates | Up to ten weeks
  Compliance is defined as number of times per week and number of hours per day of task performance
Qualitative assessment | Up to ten weeks
  Participants' reactions to the study will be gathered with Likert scale ratings of perceived problems of delivery, ease of program use, and perceived improvement of cognition. Open-ended responses to structured questions on likes and dislikes, suggestions for improvement, and overall satisfaction will also be implemented.

SECONDARY OUTCOMES:
Improvement in performance over time | Up to ten weeks
  Performance at the beginning of the training session of each task will be compared to performance at the completion of the training session of each task.
Relation of performance to mental health | At ten weeks
  Scores on pre- and post- mental health measures will also be related to task performance

CONTACTS AND LOCATIONS:
Overall Officials: Mary R Newsome, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States